CLINICAL TRIAL: NCT02435407
Title: The Sequential Oral Sensory (SOS) Intervention in Treating Children With Autism Spectrum Disorder and Limited Food Repertoire
Brief Title: The Sequential Oral Sensory Approach for Limited Food Repertoire in Children With Autism Spectrum Disorder
Acronym: SOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB file # 14-511
Record Dates: First submitted 2015-04-28; First posted 2015-05-06 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-05

CONDITIONS: Autism Spectrum Disorder; Feeding Disorder; Restricted Diet
MeSH Terms: conditions — Autism Spectrum Disorder; Feeding and Eating Disorders | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOS arm (Experimental): The Sequential Oral Sensory (SOS) approach treatment protocol, involving systematic desensitization hierarchy of skills needed to build feeding skills.
  Interventions: Behavioral: SOS
- Education arm (Active Comparator): Parents will participate in educational talks around the cause and management of feeding difficulties in children with autism spectrum disorder.
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: SOS — Ten (10) children will be randomized to participate in the SOS intervention arm. The intervention will be divided into two groups of 5 children with 2 therapists assigned. The children will attend 1 hour intervention sessions once a week for 12 weeks. Here they will be introduced to different types of foods that they would not have typically eaten in a play based group session. The SOS intervention utilizes the principle of hierarchal desensitization.
  Other Names: Sequential Oral Sensory approach
  Arms: SOS arm
Other: Education — Parents will be given three 1 hour educational talks around the aetiology and management of feeding difficulties in children with autism spectrum disorder. This will be administered at 3 distinct time points; baseline, week 6 and week 12 of the study.
  Arms: Education arm

SUMMARY:
There is a paucity of research evaluating the effectiveness of a multidisciplinary approach in an outpatient clinic setting in the management of feeding problems in children diagnosed with ASD. Current behavioural interventions geared to address this problem can be labour intensive and costly. The SOS approach for managing feeding problems in children has been adopted internationally. Thus establishing its effectiveness will be useful in providing evidenced based interventions for feeding difficulties in ASD.

DETAILED DESCRIPTION:
Feeding problems in children diagnosed with autism spectrum disorder (ASD) has been found to vary from 46-89%, with significant variability in feeding patterns. Feeding problems can lead to failure to thrive, nutritional deficiencies, growth retardation, social deficits and poor academic achievements. Common feeding problems are typified by limited food repertoire, food refusal and high frequency single food intake. The etiology of feeding problems in children with ASD is multifactorial and includes sensory issues, perseveration, avoidance of novel stimuli and food intolerance. No single aetiology has been assigned to limited food repertoire in children diagnosed with ASD. A recent meta-analysis of feeding problems and nutritional intake in children diagnosed with ASD reveals that children with ASD had more feeding problems when compared to peers (odds ratio 5.11, 95% Confidence interval (CI) 3.74-6.97). There was significantly lower intake of calcium and protein. Children diagnosed with ASD have limited food repertoire compared to typically developing children (19.0 (5.0) foods eaten vs. 22.5 (4.6) foods eaten, p value 0.0003) and they have evidence of nutritional inadequacies and poor bone growth. The impact of feeding problems extends to the home environment and may contribute to parental stress and affect bonding/ attachment of child to caregiver during mealtimes. This phenomena has not been explored in depth in current research.

Behavioural intervention using an interdisciplinary team model is the hallmark intervention for the treatment of feeding problems in children diagnosed with ASD. However there is limited research data available in this field. Behavioural intervention approaches described in the literature include stimulus control, positive reinforcement, negative reinforcement, discrimination training, extinction, punishment and desensitization. Positive reinforcement-based intervention, physical guidance, and non-removal of the spoon are techniques which have found to be useful based on case reports. These interventions require highly structured environments, are costly and at times parents are not involved in the management plan, thus limiting generalizability. There is no consensus regarding which technique is superior and more effective.

There are three published interventional studies which directly address feeding problems in ASD. These span from intensive inpatient management to behavioural patient based curriculum. A retrospective chart review of 37 children over a 2 year period seen in group intervention sessions using the Sequential Oral Sensory (SOS) approach showed some promise in increasing food variability and intake. The Sequential Oral Sensory (SOS) approach is a multidisciplinary program for assessing and treating children with feeding and weight problems. This program uses a systematic desensitization hierarchy of skills necessary for children to progress with eating various food textures. The technique is patient controlled, where the patient is "allowed to move away" from the exposure. The goal of the therapy is to maintain a competing response in the face of increasing incremental exposures. The SOS approach if effective presents a more affordable treatment option, in a natural outpatient setting and utilizes parental participation under supervision which may translate to generalizability to the home environment. Given the prevalence of feeding challenges in ASD exploring this option should be undertaken given its suggested implications.

ELIGIBILITY:
Inclusion Criteria:

* •Children diagnosed with Autism Spectrum Disorder based upon an Autism Diagnostic Observation Schedule12 (ADOS) and Diagnostic and Statistical Manual (DSM)-IV or DSM-V interview.

  * Age 48 months - 96 months
  * Child who is physically able to observe others in a group setting
  * Children identified as having limited food repertoire < 20 food in dietary repertoire
  * Test of Adaptive function: Vineland Adaptive Behavioural Scale- 2nd Edition form13
  * Child and caregiver/ parent committed to attend 12 sessions
  * Parents are fluent in English
  * Parent total Difficult Child score on the Parental Stress Index short form14 is above the 90th percentile (which is deemed clinically significant)

Exclusion Criteria:

* •A child who has an anatomical cause for feeding problems such as cleft palate or significant oromotor abnormality

  * Child diagnosed with failure to thrive
  * Child who is unable to sit at the table during mealtime
  * Child with significant motor difficulties
  * Children in foster care
  * Participation in concurrent feeding clinic/ intervention
  * Child with moderate to severe cognitive/intellectual impairment

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in the number of foods eaten after 12 weeks of intervention as determined by the 3 day food diary | 12 weeks
  The primary aim of the current proposal is to evaluate the effectiveness of the SOS Approach intervention for increasing the food repertoire in children diagnosed with ASD and limited food repertoire. A 12 week, unblinded randomized controlled trial of SOS approach intervention matched by age will be conducted. Following a screening visit, subjects assigned to the intervention group will return at baseline and then weekly for 12 weeks.

SECONDARY OUTCOMES:
Change in the level of parental stress around meal times after 12 weeks of intervention as determined by the Parent Stress Index questionnaire | 12 weeks
  The secondary study aim is to investigate if participation in the SOS approach intervention will lead to decreased parental stress around mealtime feeding
Description of the sensory profiles of participants as determined by the Short Sensory Profile- short form Questionnaire | At baseline
  To investigate the sensory profiles of subjects participating in the study.

OTHER OUTCOMES:
To determine parental satisfaction as determined by the Canadian Occupation Performance Measure | 12 weeks
  To assess parents satisfaction with their child's performance during meals after participating in the SOS intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Smile, MD, MSc., Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada